CLINICAL TRIAL: NCT04211610
Title: Troponin Excretion in Urine in Patients With and Without Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Yasmeen Abu Fraiha, Internal Medicine Resident, Internal Medicine Department B, Soroka University Medical Center
Other Study IDs: 0234-19-SOR
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Diseases; Acute Myocardial Infarction
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples Without DNA — Blood and urine samples will be collected from each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1 - Healthy subjects without any evidence of cardiac o: Inclusion criteria:
  1. Normal serum troponin (below the 99th percentile)
  2. GFR 60ml/min
  3. Proteinuria <1gr/gr creatinine
  Blood and urine samples will be collected for troponin and other measures.
  Interventions: Diagnostic Test: Blood and urine sampling
- Group 2 - Subjects with acute myocardial infarction and norm: Inclusion criteria:
  1. At least one measurements of serum troponin above the 99th percentile, with either a rise or fall in cardiac troponin levels.
  2. GFR 60ml/min/1.73m2
  Blood and urine samples will be collected for troponin and other measures.
  Interventions: Diagnostic Test: Blood and urine sampling
- Group 3 - Subjects with acute myocardial infarction and decr: Inclusion criteria - Group 3a:
  1. At least one measurements of serum troponin above the 99th percentile, with either a rise or fall in cardiac troponin levels.
  2. 30 GFR <60ml/min/1.73m2
     Inclusion criteria - Group 3b:
  3. At least one measurements of serum troponin above the 99th percentile, with either a rise or fall in cardiac troponin levels.
  4. GFR <30ml/min/1.73m2
  Blood and urine samples will be collected for troponin and other measures.
  Interventions: Diagnostic Test: Blood and urine sampling
- Group 4 - Subjects with decreased GFR but without any eviden: Inclusion criteria - Group 4a:
  1. Normal serum troponin (below the 99th percentile)
  2. No known past medical history of any cardiac disease and/or procedure.
  3. 30 GFR <60ml/min/1.73m2
     Inclusion criteria - Group 4b:
  4. Normal serum troponin (below the 99th percentile)
  5. No known past medical history of any cardiac disease and/or procedure.
  6. GFR <30ml/min/1.73m2
  Blood and urine samples will be collected for troponin and other measures.
  Interventions: Diagnostic Test: Blood and urine sampling
- Group 5 - Subjects with chronic myocardial injury and normal: Inclusion criteria:
  1. At least one measurements of serum troponin above the 99th percentile, with neither a rise nor fall in cardiac troponin levels.
  2. GFR 60ml/min/1.73m2
  Blood and urine samples will be collected for troponin and other measures.
  Interventions: Diagnostic Test: Blood and urine sampling
- Group 6 - patients on RRT: Inclusion criteria:
  a. Patients who are dependent on renal replacement therapy, including hemodialysis, peritoneal or hemodiafiltration.
  Blood and urine samples will be collected for troponin and other measures.
  Interventions: Diagnostic Test: Blood and urine sampling

INTERVENTIONS:
Diagnostic Test: Blood and urine sampling — * Blood tests - hs-cTnT, hs-cTnI, complete metabolic panel including urea, creatinine, albumin and myoglobin
  * Urine tests - hs-cTnT, hs-cTnI, urea, creatinine, albumin, total protein, β2-microglobulin.

SUMMARY:
In this study, in order to better understand the mechanism of troponin clearance and the reason for elevated troponin levels in patients with CKD, we aim to evaluate quantitatively the excretion of troponin in the urine in patients with and without CKD, and with and without myocardial injury. We will compare urinary troponin levels with blood troponin levels in these patients. In addition, we will compare the levels of hs-cTnT and hs-cTnI in the patients' sera and urine.

DETAILED DESCRIPTION:
The study population will be screened at the internal wards, the nephrology ward and clinic, and the intensive cardiac care unit (ICCU) of Soroka Medical Center. It will include patients who suffer from AMI, patients with CKD with and without any cardiac disease and patients with no known renal or cardiac disease.

The following information and measurements will be collected:

Demographics - age, sex, weight, height. Past medical history - specifically regarding renal and cardiac diseases and procedures.

Measured variables in blood serum - troponin T, troponin I, creatinine, total protein, albumin, myoglobin Measured variables in urine - troponin T, troponin I, creatinine, total protein, albumin, microalbumin, β2-microglobulin Calculations - GFR (according to MDRD equation), troponin correction to creatinine (gr troponin per gr creatinine), troponin excretion ( ), urine albumin/creatinine ratio, urine protein/creatinine ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are able to give informed consent.
2. Age ≥ 18

Exclusion Criteria:

1. Pregnant women
2. Patients after kidney transplantation.
3. Patients after heart transplantation.
4. Anuric patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be screened at the internal wards, the nephrology ward and clinic, and the intensive cardiac care unit (ICCU) of Soroka Medical Center. It will include patients who suffer from AMI, patients with CKD with and without any cardiac disease and patients with no known renal or cardiac disease. The study population will be enrolled according to the above inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Troponin T in blood vs. urine | 1 year
  Quantitative measurements of hs-cTnT in blood and urine
Troponin I in blood vs. urine | 1 year
  Quantitative measurements of hs-cTnI in blood and urine

SECONDARY OUTCOMES:
Troponin excretion in urine compared to creatinine | 1 year
  Comparing urine troponin levels to urine creatinine, albumin, β2-microglobulin
Troponin excretion in urine compared to albumin | 1 year
  Comparing urine troponin levels to urine albumin
Troponin excretion in urine compared to β2-microglobulin | 1 year
  Comparing urine troponin levels to urine β2-microglobulin

CONTACTS AND LOCATIONS:
Overall Officials: Yosef Haviv, MD, Study Chair — Soroka UMC, Nephrology Department, Director
Locations (1):
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Twerenbold R, Wildi K, Jaeger C, Gimenez MR, Reiter M, Reichlin T, Walukiewicz A, Gugala M, Krivoshei L, Marti N, Moreno Weidmann Z, Hillinger P, Puelacher C, Rentsch K, Honegger U, Schumacher C, Zurbriggen F, Freese M, Stelzig C, Campodarve I, Bassetti S, Osswald S, Mueller C. Optimal Cutoff Levels of More Sensitive Cardiac Troponin Assays for the Early Diagnosis of Myocardial Infarction in Patients With Renal Dysfunction. Circulation. 2015 Jun 9;131(23):2041-50. doi: 10.1161/CIRCULATIONAHA.114.014245. Epub 2015 May 6. PMID 25948542
- [Background] Freda BJ, Tang WH, Van Lente F, Peacock WF, Francis GS. Cardiac troponins in renal insufficiency: review and clinical implications. J Am Coll Cardiol. 2002 Dec 18;40(12):2065-71. doi: 10.1016/s0735-1097(02)02608-6. PMID 12505215
- [Background] Kanderian AS, Francis GS. Cardiac troponins and chronic kidney disease. Kidney Int. 2006 Apr;69(7):1112-4. doi: 10.1038/sj.ki.5000174. PMID 16531987
- [Background] Ziebig R, Lun A, Hocher B, Priem F, Altermann C, Asmus G, Kern H, Krause R, Lorenz B, Mobes R, Sinha P. Renal elimination of troponin T and troponin I. Clin Chem. 2003 Jul;49(7):1191-3. doi: 10.1373/49.7.1191. No abstract available. PMID 12816921
- [Background] Petra, P., Tomo, S., Ingrid, P., Jurica, V., Andrea, R., & Sonja, P. Urine Concentrations of High-Sensitivity Cardiac Troponin I in Healthy Adults - Preliminary Reference Intervals. Acta Med Croatica , 461-465, 2018
- [Background] Petra, P., Tomo, S., Ingrid, P., Ana, S., Matija, B., & Sonja, P. Urine High-Sensitive Troponin I Measuring in Patients with Hypertension. Signa Vitae , 13(SUPPL 3): 62-64, 2017
- [Background] Friden V, Starnberg K, Muslimovic A, Ricksten SE, Bjurman C, Forsgard N, Wickman A, Hammarsten O. Clearance of cardiac troponin T with and without kidney function. Clin Biochem. 2017 Jun;50(9):468-474. doi: 10.1016/j.clinbiochem.2017.02.007. Epub 2017 Feb 11. PMID 28193484
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Glob Heart. 2018 Dec;13(4):305-338. doi: 10.1016/j.gheart.2018.08.004. Epub 2018 Aug 25. No abstract available. PMID 30154043
- [Background] Dubin RF, Li Y, He J, Jaar BG, Kallem R, Lash JP, Makos G, Rosas SE, Soliman EZ, Townsend RR, Yang W, Go AS, Keane M, Defilippi C, Mishra R, Wolf M, Shlipak MG; CRIC Study Investigators. Predictors of high sensitivity cardiac troponin T in chronic kidney disease patients: a cross-sectional study in the chronic renal insufficiency cohort (CRIC). BMC Nephrol. 2013 Oct 22;14:229. doi: 10.1186/1471-2369-14-229. PMID 24148285